CLINICAL TRIAL: NCT03206164
Title: HealthMatters@24/7 Asynchronous Health Promotion eLearning for People Supporting Adults With Intellectual and Developmental Disabilities
Brief Title: HealthMatters@24/7 eLearning for People Supporting Adults With Intellectual and Developmental Disabilities
Acronym: HM@24/7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Beth Marks, Research Associate Professor, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0754; P30AG022849 (NIH); UL1TR002003 (NIH)
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Obesity; Hypertension; Hypercholesterolemia; Hyperglycemia
Keywords: Health Services Research
MeSH Terms: conditions — Obesity; Hypertension; Hypercholesterolemia; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Methods: We will convert the evidence based HealthMatters Train the Trainer Workshop for Instructors, synchronous, live webinar training course into HealthMatters@24/7, an asynchronous, e-learning training course for staff to plan, conduct, and evaluate the HealthMatters Program for people with IDD in residential and day/employment community-based organizations (CBOs).
  Design. We will utilize a two-group (Table 1) pre-test/post test quasi-experimental design wherein the Experimental Group will receive HealthMatters@24/7 training and the Control Group will receive the customary real-time (live) webinar training (HealthMatters Train the Trainer Workshop).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asynchronous, eLearning Intervention (Experimental): Participants in the asynchronous, eLearning Intervention Group will participate in the on-demand HealthMatters Program Instructor Training Course that will be continuously and readily available.
  Interventions: Other: Asynchronous, eLearning Intervention
- Synchronous, Live Webinar Comparison (Active Comparator): Participants in the synchronous, Live Webinar Comparison Group will receive HealthMatters Program Instructor Training Course via a live instructor taught 3-part live webinar.
  Interventions: Other: Asynchronous, eLearning Intervention

INTERVENTIONS:
Other: Asynchronous, eLearning Intervention — 20 CBOs with 3-member team (n= 30) will be recruited and placed into either the experimental or the comparison group.

SUMMARY:
The barriers faced by people with intellectual and developmental disabilities (IDD) begin in their mid to late 20s and often mirror the experiences of older adults (50+) living in the U.S. While evidence for successful population-specific health promotion programs and training, such as the 12-Week HealthMatters Program has been documented, an urgent need exists for continuous, readily available, on-demand training in these programs. Online training can substantially aid the widespread translation of evidence-based programs into practice and policy. This proposal seeks to test the effectiveness of an enhanced mode of translating the HealthMatters program into practice through the use of an on-demand e-Learning platform (HealthMatters@24/7) for staff in community based organizations (CBOs) in one state; thereby advancing the science of translational research. HO1. More CBOs in the asynchronous training program will have developed Strategic Action Plans for Health and Wellness, established Wellness Committees, and have equal or more resources and improved culture for health promotion at 1 year compared to CBOs participating in the current live HealthMatters TtT Workshop webinar. HO2. Staff in the asynchronous training group will have improved levels of learner/instructor satisfaction (job productivity, job performance, job satisfaction, organizational commitment, convenience) toward the training immediately after completing the enhanced mode of training, HM@24/7 compared to staff trained using the current live HealthMatters TtT Workshop webinar.

DETAILED DESCRIPTION:
The barriers faced by people with intellectual and developmental disabilities (IDD) begin in their mid to late 20s and often mirror the experiences of older adults (50+) living in the U.S. While evidence for successful population-specific health promotion programs and training, such as the 12-Week HealthMatters Program has been documented, an urgent need exists for continuous, readily available, on-demand training in these programs. Online training can substantially aid the widespread translation of evidence-based programs into practice and policy. Consistent with the mission of the Midwest Roybal Center for Health Promotion and Translation, our proposed study, HealthMatters@24/7 eLearning, is guided by the RE-AIM framework to evaluate the reach, efficacy, adoption, implementation, and maintenance of the HealthMatters Program for maximal positive impact on the health of people with IDD. The goal of HealthMatters@24/7 eLearning is to develop a low cost, readily accessible comprehensive staff training that will improve staff job performance, satisfaction, and organizational commitment to the provision of health friendly services while creating a productive and competitive workforce. These conditions will enable more community-based organizations to offer the program efficiently, thereby increasing access to HealthMatters among older adults with IDD.

ELIGIBILITY:
Inclusion Criteria:

* Must work in a community based organization providing services to people with intellectual and developmental disabilities
* Must read english
* Must be over the age of 18

Exclusion Criteria:

* Do not work in a community based organization providing services to people with intellectual and developmental disabilities
* Do not read english
* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
online organizational HealthMatters Assessments (oHMA) | 1 year
  oHMA evaluates organizational needs and capacity for developing a health promotion plan including programs, services, environmental support, resources, and culture to provide health promoting activities.

SECONDARY OUTCOMES:
Process Evaluation | 3 months
  Will evaluate participants ability to develop and implement Strategic Action Plans for Health and Wellness, Wellness Committees, and greater numbers of organizational resources for health promotion
36-item Corporate eLearning Survey | 1 year
  Measures participants perception of on-job productivity, job performance, job satisfaction and organizational commitment.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Marks, PhD, RN, Study Director — Research Associate Professor
Locations (1):
- UIC, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heller T, Fisher D, Marks B, Hsieh K. Interventions to promote health: crossing networks of intellectual and developmental disabilities and aging. Disabil Health J. 2014 Jan;7(1 Suppl):S24-32. doi: 10.1016/j.dhjo.2013.06.001. PMID 24456681
- [Background] Anderson LL, Humphries K, McDermott S, Marks B, Sisirak J, Larson S. The state of the science of health and wellness for adults with intellectual and developmental disabilities. Intellect Dev Disabil. 2013 Oct;51(5):385-98. doi: 10.1352/1934-9556-51.5.385. PMID 24303825
- [Background] Marks B, Sisirak J, Chang YC. Efficacy of the HealthMatters program train-the-trainer model. J Appl Res Intellect Disabil. 2013 Jul;26(4):319-34. doi: 10.1111/jar.12045. Epub 2013 Apr 16. PMID 23589506
- [Background] Heller T, Hsieh K, Rimmer JH. Attitudinal and psychosocial outcomes of a fitness and health education program on adults with down syndrome. Am J Ment Retard. 2004 Mar;109(2):175-85. doi: 10.1352/0895-8017(2004)1092.0.CO;2. PMID 15000672
- [Background] Scott HM, Havercamp SM. Systematic Review of Health Promotion Programs Focused on Behavioral Changes for People With Intellectual Disability. Intellect Dev Disabil. 2016 Feb;54(1):63-76. doi: 10.1352/1934-9556-54.1.63. PMID 26824134
- [Background] Rimmer JH, Yamaki K, Davis BM, Wang E, Vogel LC. Obesity and overweight prevalence among adolescents with disabilities. Prev Chronic Dis. 2011 Mar;8(2):A41. Epub 2011 Feb 15. PMID 21324255
- [Background] Zontek TL, Isernhagen JC, Ogle BR. Psychosocial factors contributing to occupational injuries among direct care workers. AAOHN J. 2009 Aug;57(8):338-47. doi: 10.3928/08910162-20090716-03. PMID 19650606
- [Background] Ellis, P.F. and K.D. Kuznia, Corporate Elearning Impact on Employees. Global Journal of Business Research, 2014. 8(4): p. 1 - 15.
- [Background] Marks, B., J. Sisirak, and T. Heller, Health Matters: The Exercise and Nutrition Health Education Curriculum for Adults with Developmental Disabilities. 2010, Philadelphia: Brookes Publishing.
- See also: Website for the HealthMatters Program — http://healthmattersprogram.org

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT03206164/Prot_SAP_000.pdf